CLINICAL TRIAL: NCT03389646
Title: CERAMENTTM|G and V in the Management of Hip and Knee Arthroplasty Revisions (Revision Arthroplasty Italy)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RAI2017
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Hip Prosthesis Infection; Knee Prosthesis Infection

STUDY DESIGN:
Intervention Model Description: Prospective with retrospective matched controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated with Device: Including sham (Active Comparator): Treated with CERAMENTTM|G or V for filling of bone defects in the tibia and/or femur and/or the acetabulum.
  Interventions: Device: CERAMENT G V
- Control (No Intervention): Control without CERAMENT device

INTERVENTIONS:
Device: CERAMENT G V — During the removal of hip and knee prostheses usually bone defects occur at the intramedullary canal of the tibia and or / femur and /or acetabulum. These bone defects are filled with CERAMENTTM|G or V during the re-implantation of the cementless or hybrid revision THA or TKA. CERAMENTTM|G or V can be directly injected into the intramedullary canal or bone defect at the acetabulum. Alternatively and preferably, the surface of the prostheses shafts can be used to transfer CERAMENTTM|G or V into the bone defects. For information of handling and mixing please see the attached instructions for use (IFU).
  Arms: Treated with Device: Including sham

SUMMARY:
Open-label, multicentre, prospective cohort, observational clinical trial with a retrospective control group to evaluate the effectiveness and safety of CERAMENTTM| G or V used for filling of bone defects in the tibia and / or femur shaft and/or acetabulum in patients scheduled for two-stage hip or knee prosthesis re-implantation for PJI or aseptic loosening.

The results will be compared to a cohort of patients, which have been treated before the introduction of CERAMENTTM|G or V for the same indication.

Due to the observational character of the study, there will be no patient randomization and the clinicians in the study will remain entirely free to decide on the treatment of the patients according to established clinical practice.

Only patients for whom therapeutic strategy for the use of the product for filling bone defects is already planned according to local clinical practice, at the time of informed consent form signature, will be enrolled in this study. Thus, the decision for the choice of the surgical treatment, will not be influenced by the inclusion of the patient in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study related procedure.
2. Male or female age ≥ 18 and ≤ 85 years.
3. Patients diagnosed with aseptic prosthetic loosening and scheduled for a one-stage hip or knee cementless or hybrid revision prosthesis implantation
4. Patients with an interval spacer and scheduled for hip or knee cementless or hybrid revision prosthesis implantation.
5. For those patients with an interval spacer, previous infection caused by microorganism(s) sensitive to gentamicin or vancomycin.
6. Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

1. Unable to give written informed consent.
2. Medically unfit for operative intervention.
3. Soft-tissue defects that prevent direct skin closure at revision surgery.
4. Females who are pregnant or lactating.
5. Females of child bearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of child bearing potential taking acceptable contraceptive precautions may be included.
6. Known allergy to gentamicin or vancomycin (or related antibiotics).
7. Patients with previous nephro- or ototoxicity events due to aminoglycoside and/or vancomycin (or glycopeptides) use.
8. Presence of relevant contraindications as described in the EU CE mark Instructions for Use (IFU).
9. Myasthenia gravis.
10. Need of a fully cemented joint prosthesis.
11. Psychiatric or neurological disorders.
12. Active infection at the site of surgery as diagnosed by clinical and/or laboratory and/or imaging investigations.

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-09-27 (Estimated); Study Completion 2019-09-27 (Estimated)

PRIMARY OUTCOMES:
incidence of post-surgical infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: CARLO L ROMANO, MD, Principal Investigator — IRCCS GALEAZZI
Locations (1):
- Irccs Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No